CLINICAL TRIAL: NCT01696149
Title: The Effects of High and Low Frequency Transcutaneous Electrical Nerve Stimulation on Sympathetic Skin Response and Skin Temperature
Brief Title: Effects of High and Low Frequency TENS on Sympathetic Skin Response and Skin Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, samaneh ebrahimi, PhD candidate, Shiraz University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 87-4520
Record Dates: First submitted 2012-09-18; First posted 2012-09-28 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Effects of TENS on Sympathetic Skin Response
Keywords: TENS, sympathetic skin response, skin temperature
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- electrical nerve stimulation (Experimental): All subjects participated, randomly, in a 4 Hz transcutaneous electrical nerve stimulation session, a 110 Hz transcutaneous electrical nerve stimulation session, and a control (off-transcutaneous electrical nerve stimulation) session. Each session consisted of a 20- minute stimulation period and a 10-minute follow up period
  Interventions: Device: transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation — All subjects participated, randomly, in a 4 Hz TENS session, a 110 Hz TENS session, and a control (off-TENS) session. Each session consisted of a 20- minute stimulation period and a 10-minute follow up period.
  Other Names: TENS

SUMMARY:
The aim of this study was to determine the effects of 4 Hz and 110 Hz transcutaneous electrical nerve stimulation on the sympathetic nervous system via measuring the sympathetic skin response (SSR) and skin temperature.

DETAILED DESCRIPTION:
15 healthy subjects (8 females, 7 males) with a mean age of 22.6 ± 3.7 years participated in this study.

All subjects participated, randomly, in a 4 Hz TENS session, a 110 Hz TENS session, and a control (off-TENS) session. Each session consisted of a 20- minute stimulation period and a 10-minute follow up period.

Outcome measures: Sympathetic skin response from the simulated (Right) hand and skin temperature of both stimulated (Right) and none stimulated (Left) hand was measured 15 seconds before, just 15 seconds after, and 10 minutes after application of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 30 years

Exclusion Criteria:

* History of cardiovascular, neurologic or musculoskeletal disease
* Taking medication at the time of the study

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Changes of sympathetic skin response | 15 seconds before, just 15 seconds after, and 10 minutes after application of interventions
  Sympathetic skin response from the simulated (Right) hand was measured 15 seconds before, just 15 seconds after, and 10 minutes after application of interventions.

SECONDARY OUTCOMES:
Changes of skin temperature | 15 seconds before, just 15 seconds after, and 10 minutes after application of interventions
  skin temperature of both stimulated (Right) and none stimulated (Left) hand was measured 15 seconds before, just 15 seconds after, and 10 minutes after application of interventions

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh Dehghan, Principal Investigator — Shiraz University of Medical Sciences